CLINICAL TRIAL: NCT04049058
Title: Evaluation of Quality of Life After Orthognathic Surgery in a Cleft Lip and Palate Context
Acronym: ORTHOQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_55; 2018-A03376-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Palate, Cleft
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare, prospectively, the quality of life of patients with cleft lip and palate before and after orthognathic surgery. This is done through two validated questionnaires: OHIP-14 (Oral Health Impact Profile) and OQLQ (Orthognathic Quality of Life Questionnaire) Improving the quality of life is the goal of any functional treatment. The demonstration of its improvement would validate the validity of this additional surgery for patients with cleft lip and palate.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman ; Age: adolescents (12-17 years) and adults; Specific medical conditions: cleft lip and palate, malocclusion
* Non-opposition of the patient
* Patient willing to comply with all procedures of the study and its duration

Exclusion Criteria

* Cancellation of orthognathic surgery
* Impossibility to receive enlightened information, impossibility to participate in the totality of the study, impossibility to complete only the questionnaire

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cleft lip and palate with malocclusion and indication of orthognathic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change of the OQLQ (Orthognathic Quality of Life Questionnaire) questionnaire score between the preoperative assessment and at 6 months postoperatively. | between the preoperative assessment and at 6 months postoperatively.
  The OQLQ questionnaire is composed of 22 items that can be rated from 0 to 4. The score varies from 0 to 88. This questionnaire is specific to the evaluation of quality of life in relation to orthognathic surgery.

SECONDARY OUTCOMES:
Change of OHIP-14 questionnaire score (Oral Health Impact Profile) between preoperative evaluation and at 6 months postoperatively. | between the preoperative assessment and at 6 months postoperatively.
  The questionnaire is a non-specific questionnaire assessing quality of life in relation to general oral health. It is composed of 14 questions that can be scored from 0 to 4. The score varies from 0 to 56.
Change of OQLQ (Orthognathic Quality of Life Questionnaire) by type of orthognathic surgery | at 6 months
  the type of orthognathic surgery performed = monomaxillary versus bimaxillary
Change of OHIP-14 (Oral Health Impact Profile) by type of orthognathic surgery | at 6 months
  the type of orthognathic surgery performed = monomaxillary versus bimaxillary

CONTACTS AND LOCATIONS:
Overall Officials: Romain Nicot, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France